CLINICAL TRIAL: NCT03191071
Title: Procalcitonin and Lung Ultrasonography Point-of-care Testing to Decide on Antibiotic Prescription in Patients With Lower Respiratory Tract Infection at Primary Care Level: Pragmatic Cluster Randomized Trial
Brief Title: An Algorithm to Decide on Antibiotic Prescription in Lower Respiratory Tract Infection in Primary Care
Acronym: UltraPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr Boillat-Blanco Noemie, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SNF 407240_167133/1
Record Dates: First submitted 2017-05-21; First posted 2017-06-19 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Lower Resp Tract Infection
Keywords: pneumonia; procalcitonin; lung ultrasound; point of care testing; antibiotic prescription; respiratory pathogens; host biomarkers
MeSH Terms: conditions — Pneumonia | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Randomized clustered pragmatic trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- UltraPro (Experimental): General practitioners randomly assigned to the UltraPro arm will be responsible to recruit patients fulfilling the inclusion criteria and manage them using the UltraPro algorithm.
  The UltraPro algorithm combines the result of a procalcitonin point-of-care test with lung ultrasound result to decide on antibiotic prescription. Blood sampling will be performed to identify potential novel biomarkers. Naso-pharyngeal swabs as well as sputum culture will allow for microbiologic identification of aetiological agents.
  Interventions: Diagnostic Test: UltraPro; Diagnostic Test: Blood sampling; Diagnostic Test: Naso-pharyngeal swab and sputum culture
- Procalcitonin (Experimental): General practitioners randomly assigned to the procalcitonin arm will be responsible to recruit patients fulfilling the inclusion criteria and manage them using the procalcitonin algorithm.
  The procalcitonin point-of-care test will be performed, as described above, to decide on antibiotic prescription. Blood sampling will be performed to identify potential novel biomarkers. Naso-pharyngeal swabs as well as sputum culture will allow for microbiologic identification of aetiological agents.
  Interventions: Diagnostic Test: Procalcitonin; Diagnostic Test: Blood sampling; Diagnostic Test: Naso-pharyngeal swab and sputum culture
- Usual Care (Active Comparator): General practitioners randomly assigned to the usual care arm will be responsible to recruit patients fulfilling the inclusion criteria and will manage and treat these patients as they usually do. Only general practitioners who do not use procalcitonin and lung ultrasonography routinely will be included in the usual care arm.
  Naso-pharyngeal swabs as well as sputum culture will be performed to allow for microbiologic identification of aetiological agents.
  Interventions: Diagnostic Test: Naso-pharyngeal swab and sputum culture

INTERVENTIONS:
Diagnostic Test: UltraPro — First, procalcitonin will be measured using a rapid point-of-care test. In case of elevated procalcitonin result (≥0.25 µg/L), a lung ultrasound will be performed to look for the presence of a lung infiltrate or consolidation suggesting the presence of community acquired pneumonia. A portable ultrasound machine with a convex probe, that will be provided to the general practitioner by the study, will be used.
  The lung ultrasound will be done following international evidence-based recommendations for point-of-care lung ultrasound using the basic eight-region sonographic technique and the criteria for positive scan and positive examination for the diagnosis of pneumonia .
  Arms: UltraPro
Diagnostic Test: Procalcitonin — Procalcitonin will be measured using a rapid point-of-care test
  Arms: Procalcitonin
Diagnostic Test: Blood sampling — A venous blood sample (17.5 mL) will be collected. Whole blood and plasma will be stored at - 80°C. Further analysis will be performed in order to identify novel biomarkers and gene transcription patterns that could predict the necessity of antibiotic prescription or the severity of disease.
  Arms: Procalcitonin; UltraPro
Diagnostic Test: Naso-pharyngeal swab and sputum culture — A pooled nasal swab will be performed and sputum will be collected. Samples will be stored at -80°C. Further analysis of the naso-pharyngeal swab and cultures of sputum will be performed to identify by molecular techniques pathogens implicated in the clinical presentation.

SUMMARY:
The study is randomized clustered pragmatic trial whose objective is to decrease unnecessary antibiotic prescription in adult patients with lower respiratory tract infection managed at primary care level in Switzerland, using a simple algorithm based on 2 point of care test results

DETAILED DESCRIPTION:
The study will have two distinct phases:

The first phase will test the feasibility of the intervention (UltraPro) along a pilot study. Following the setup of a lung ultrasound training curriculum for general practitioners, the practicality of the whole UltraPro algorithm will be evaluated at primary care level.

The second phase will be a pragmatic randomized three-arm intervention study using an algorithm based on the results of procalcitonin and lung ultrasound to manage patients with lower respiratory tract infections at primary care level. The procalcitonin-ultrasound algorithm will be compared to procalcitonin-guided management alone and usual care.

ELIGIBILITY:
All patients presenting to a participating GP's office for a consultation for an acute respiratory infection (ARI) will be screened for inclusion in the study

Inclusion Criteria:

* Informed Consent as documented by signature (Informed Consent Form)
* Patients aged 18 years or more
* No antibiotics prescribed for the current episode
* Acute cough of up to 21 days duration and at least one of the following symptom or sign:
* History of fever for more than 4 days
* dyspnoea
* tachypnoea (≥ 22 cycles per minutes)
* abnormal focal finding during auscultation

Exclusion Criteria:

* Previous prescription of antibiotics for the current episode
* Working diagnosis of acute sinusitis or a non-infective disorder
* Cystic fibrosis
* Previous episode of chronic obstructive pulmonary disease exacerbation treated with antibiotics during the last 6 months
* Known pregnancy
* Severe immunodeficiency (untreated HIV infection with CD4 count < 200 cells/mm3, solid organ transplant receiver, neutropenia, treatment with corticosteroids with dose equivalent to 20 mg prednisone/day for > 28
* Admission of the patient
* GP not available for performing study
* Patient unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients prescribed an antibiotic in each arm | Assessed at day 28 after baseline
  For each arm, we will assess the proportion of patient's prescribed an antibiotic following the consultation with the general practitioner. This will be done by recording the prescription decision of the general practitioner.

SECONDARY OUTCOMES:
Duration of the episode | Assessed at day 28 after baseline
  Number of days, within the first 28 days after enrolment, during which the patient's daily activities (work or recreation) were restricted by the lower respiratory tract infection. This will be assessed by telephone follow-up consultations
Clinical failure | Day 7 after baseline
  Presence of symptoms of an ongoing or relapsing lower respiratory tract infection at 28 days after enrolment. This will be assessed by a telephone follow-up consultation.
Number of medical visits | Day 7 and Day 28 after baseline
  The incidence of supplementary medical visits for the episode of lower respiratory tract infection within 28 days of enrolment will be assessed by reporting from the general practitioners and telephone follow-up consultations
Serious adverse outcome | During the first 28 days following baseline
  Secondary hospitalisation or death of any cause or disease specific complications (lung abscess, empyema and acute respiratory distress), within 28 days of enrolment. Assessed by serious adverse event reporting, general practitioner reporting and telephone follow-up.
Duration of algorithm completion | Assessed at baseline (Day 0)
  Median duration of time spent for the medical consultation, procalcitonin testing, lung ultrasound and total time spent in the practice. These will be assessed by the general practitioner by filling in a case report form at baseline.
Satisfaction of providers | Assessed at baseline
  The overall satisfaction of general practitioners regarding the process of the consultation and its different components will be assessed using a Likert scale.
Satisfaction of patients | Assessed at day 7
  The overall satisfaction of patients regarding the process of the consultation and of follow-up will be assessed using a Likert scale. These will be assessed by telephone follow-up.
Cost / effectiveness ratio | Assessed one month after data collection is complete
  Cost / effectiveness ratio expressed as the cost required per 1% decrease of the rate of antibiotic prescription during the studio will be assessed using review of the medical records and estimation of the costs of the various process of the diagnostic algorithm based on the Swiss Federal HealthCare Law.
Aetiology of LRTIs in primary care | Assessed within the first year after data collection is complete
  Prevalence of different respiratory pathogens as assessed by realtime multiplex PCR performed on a naso-pharyngeal swab and in sputum
Host biomarkers | Assessed within the first year after data collection is complete
  Sensitivity and specificity of combinations of host biomarkers to identify patients with clinical failure or with pneumonia
Transcription patterns | Assessed within the first year after data collection is complete
  Association between SNPs in genes involved in microvascular integrity and poor outcome or clinical failure

CONTACTS AND LOCATIONS:
Overall Officials: Noémie Boillat, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Only coded and anonymous data will be made available to protect patients right to privacy

REFERENCES:
- [Derived] Geis D, Canova N, Lhopitallier L, Kronenberg A, Meuwly JY, Senn N, Mueller Y, Fasseur F, Boillat-Blanco N. Exploration of the Acceptance of the Use of Procalcitonin Point-of-Care Testing and Lung Ultrasonography by General Practitioners to Decide on Antibiotic Prescriptions for Lower Respiratory Infections: A Qualitative Study. BMJ Open. 2023 May 11;13(5):e063922. doi: 10.1136/bmjopen-2022-063922. PMID 37169498
- [Derived] Lhopitallier L, Kronenberg A, Meuwly JY, Locatelli I, Mueller Y, Senn N, D'Acremont V, Boillat-Blanco N. Procalcitonin and lung ultrasonography point-of-care testing to determine antibiotic prescription in patients with lower respiratory tract infection in primary care: pragmatic cluster randomised trial. BMJ. 2021 Sep 21;374:n2132. doi: 10.1136/bmj.n2132. PMID 34548312
- [Derived] Lhopitallier L, Kronenberg A, Meuwly JY, Locatelli I, Dubois J, Marti J, Mueller Y, Senn N, D'Acremont V, Boillat-Blanco N. Procalcitonin and lung ultrasonography point-of-care testing to decide on antibiotic prescription in patients with lower respiratory tract infection in primary care: protocol of a pragmatic cluster randomized trial. BMC Pulm Med. 2019 Aug 6;19(1):143. doi: 10.1186/s12890-019-0898-3. PMID 31387559

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT03191071/Prot_SAP_000.pdf